CLINICAL TRIAL: NCT06590571
Title: Comparison of a Pressure-controlled Hemostatic Device With Conventional Compression for Transradial Coronary Angiography and Intervention: A Prospective, Multicenter, Randomized, Controlled Trial
Brief Title: The Study for Evaluate of Satety and Dfficacy of Hemostatic Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The company stopped manufacturing the product
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Min Ku Chon, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TRAcelet study
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Percutaneous coronary intervention; Hemostasis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Simple randomization was performed at the end of each coronary angiography procedure using a randomization table provided by the website (http://stattrek.com/Tables/Random.aspx). Investigators were able to identify the assignment only after the coronary angiography procedure and before the removal of the sheath catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAcelet™ compression group (Experimental): the group using TRAcelet™ received 2 hours and 15 minutes of compression from the device with 13 cc of air being blown in, followed by 3 stepwise releases every 15 minutes through counterclockwise rotation of the dial without extracting air using a syringe. This achieved the same 3 hours of compression. The dial started at the triangle position and was set to nine, six, and three at every stepwise decompression. After three hours, the device was released.
  Interventions: Device: TRAcelet™
- Conventional compression group (Other): Patients who were assigned to the conventional group received radial artery compression by a gauze pad folded into a cuboid shape, fastened with 3M™ Durapore™ surgical tape. The gauze pad was not impregnated with prothrombotic material. Compression was released at 3 hours to check for complications. An additional one hour of compression was applied when incomplete hemostasis or hematoma was identified.
  Interventions: Other: Gauze pad

INTERVENTIONS:
Device: TRAcelet™ — The group using TRAcelet™ after transradial angiography/intervention receives 2 hours and 15 minutes of compression from the device, followed by 3 stepwise releases every 15 minutes. There are two sizes of TRAcelet™ available, large and medium. Assuming that a Korean adult's wrist size is smaller than that of the Western population, we used a medium-sized TRAcelet™.
  Arms: TRAcelet™ compression group
Other: Gauze pad — Patients received radial artery compression by a gauze pad fastened with 3M™ Durapore™ surgical tape. An additional one hour of compression was applied when incomplete hemostasis or hematoma was identified.
  Arms: Conventional compression group

SUMMARY:
The goal of this clinical trial is to compare the new pneumatic compression device TRAcelet with conventional compression method in patients undergone transradial coronary angiography. The main question it aims to answer is the achievement of successful hemostasis at 3 hours.

Researchers will compare conventional compression to see if new pneumatic device can provide better hemostasis.

DETAILED DESCRIPTION:
Although there are several devices available for radial artery hemostasis, conventional compression with a gauze pad is thought to be the easiest method. One of the devices with a pneumatic compression balloon is the TRAcelet™, and there is not much research comparing the device and conventional compression method. Therefore, the investigators aimed to compare the pneumatic compression device TRAcelet with the conventional compression method in patients who underwent transradial coronary angiography/intervention.

The primary endpoint was the achievement of successful hemostasis at 3 hours. Successful hemostasis was defined as the absence of oozing and the absence of hematoma formation after the device was released. If incomplete hemostasis was observed after 3 hours, the achievement of hemostasis after an additional hour of compression was also considered successful. Conversely, if hemostasis could not be established, it was defined as unsuccessful hemostasis. The secondary endpoints included the total banding time, local vascular complications classified according to the EASY (Early Discharge After Transradial Stenting of Coronary Arteries) scale, pain or discomfort related to the transradial approach, which was assessed by the participants using the Wong-Baker Faces Pain Rating Scale and numeric pain rating scale, and the RAO at one month.

ELIGIBILITY:
Inclusion Criteria:

* aged over 20 years
* Underwent coronary angiography under suspicion of coronary artery disease
* Agreed to participate in the trial before the coronary angiography procedure

Exclusion Criteria:

* Bleeding tendency due to congenital or acquired disorders such as severe liver disease, thrombocytopenia (platelet count below 50,000 cells/μL)
* Those who were on anticoagulants.
* Patients who could not provide voluntary consent.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The achievement of successful hemostasis at 3 hours. | 3 hours after the procedure
  Successful hemostasis was defined as the absence of oozing and the absence of hematoma formation after the device was released. If incomplete hemostasis was observed after 3 hours, the achievement of hemostasis after an additional hour of compression was also considered successful.

SECONDARY OUTCOMES:
total hemostasis time | 4 hours after the procedure
  Total banding time
complication of procedures | 2 hours after the procedure
  Vascular complications occurring after 2 hours of compression hemostasis at the procedure site
complication of procedures | One month after the procedure
  Radial artery occlusion
complication of procedures | 4 hours after the procedure
  Pain assessment : numeric pain scale(The Numeric Pain Scale is a tool used to assess a person level of pain. It typically involves asking the patient to rate their pain on a scale from 0 to 10)
complication of procedures | 4 hours after the procedure
  Pain assessment :Wong-Baker Facial Grimace Scale(The Wong-Baker Facial Grimace Scale is a tool used to assess pain in patients who may have difficulty verbalizing their pain, such as children or individuals with cognitive impairments. It involves a series of facial expressions that represent varying levels of pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsannam-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The data used to support the findings of this study are available from the corresponding author upon request.
Supporting Information: Study Protocol, SAP
Time Frame: For about an year.